CLINICAL TRIAL: NCT00409175
Title: Safety and Efficacy of Orally Administered Fx-1006A in Patients With Familial Amyloid Polyneuropathy (FAP): A Randomized, Double-blind, Placebo-controlled Study
Brief Title: Safety and Efficacy Study of Fx-1006A in Patients With Familial Amyloidosis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FX-005; B3461020
Record Dates: First submitted 2006-12-06; First posted 2006-12-08 (Estimated); Results first posted 2012-12-17 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-11

CONDITIONS: Familial Amyloid Polyneuropathy
Keywords: FAP; Fx-1006A; transthyretin; TTR; amyloid; polyneuropathy; V30M; familial; hereditary; amyloidosis; FoldRx
MeSH Terms: conditions — Amyloid Neuropathies, Familial; Alzheimer Disease; Polyneuropathies; Amyloidosis | interventions — tafamidis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1. (Experimental): Fx-1006A
  Interventions: Drug: Fx-1006A
- 2. (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fx-1006A — Fx-1006A 20mg or matched placebo once daily (at the same time each day) for a period of 18 Months
  Arms: 1.
Drug: Placebo — Fx-1006A 20mg or matched placebo once daily (at the same time each day) for a period of 18 Months
  Arms: 2.

SUMMARY:
This study will examine whether Fx-1006A is effective in halting the progression of Familial Amyloid Polyneuropathy (FAP).

Deposition of TTR amyloid is associated with a variety of human diseases. Deposition of amyloid fibrils of variant TTR (primarily V30M) in peripheral nerve tissue produces the condition called FAP.

The prevention of the formation of amyloid by stabilization of the TTR native state should constitute an effective therapy for amyloid diseases. Therapeutic intervention with a TTR stabilizer drug, such as Fx-1006A, is hypothesized to stop progression of the disease in FAP patients. FAP is a uniformly fatal disease and Fx-1006A is intended to halt the relentless neurological deterioration FAP patients experience.

This Phase 2/3 study will enroll early to mid-stage FAP patients in order to interrupt and stabilize the disease at a point in time where progression of motor and autonomic dysfunction can be maximally effected. Male and female patients with FAP with documented V30M TTR mutation will receive Fx-1006A or placebo once daily for a period of eighteen (18) months.

DETAILED DESCRIPTION:
Deposition of TTR amyloid is associated with a variety of human diseases. Deposition of amyloid fibrils of variant TTR (primarily V30M) in peripheral nerve tissue produces the condition called FAP.

The prevention of the formation of amyloid by stabilization of the TTR native state should constitute an effective therapy for amyloid diseases. Therapeutic intervention with a TTR stabilizer drug, such as Fx-1006A, is hypothesized to stop progression of the disease in FAP patients. FAP is a uniformly fatal disease and Fx-1006A is intended to halt the relentless neurological deterioration FAP patients experience.

This Phase 2/3 study will enroll early to mid-stage FAP patients in order to interrupt and stabilize the disease at a point in time where progression of motor and autonomic dysfunction can be maximally effected. Male and female patients with FAP with documented V30M TTR mutation will receive Fx-1006A or placebo once daily for a period of eighteen (18) months.

ELIGIBILITY:
Inclusion Criteria:

1. Amyloid documented by biopsy.
2. Documented V30M TTR mutation.
3. Peripheral and/or autonomic neuropathy with a Karnofsky Performance Status ≥50.
4. Patient is 18-75 years old.
5. If female, patient is post-menopausal, surgically sterilized, or willing to use an acceptable method of birth control. If male with a female partner of childbearing potential, willing to use an acceptable method of birth control for the duration of the study. For both females and males, birth control must be used for at least 3 months after the last dose of study medication.
6. Patient is, in the opinion of the investigator, willing and able to comply with the study medication regimen and all other study requirements.

Exclusion Criteria:

1. Chronic use of non-steroidal anti-inflammatory drugs (NSAIDs).
2. Primary amyloidosis.
3. If female, patient is pregnant or breast feeding.
4. Prior liver transplantation.
5. No recordable sensory threshold for vibration perception in both feet, as measured by CASE IV.
6. Positive results for hepatitis B surface antigen (HBsAg), anti-hepatitis C virus (HCV), and/or human immunodeficiency virus (HIV).
7. Renal insufficiency or liver function test abnormalities.
8. New York Heart Association (NYHA) Functional Classification ≥III.
9. Other causes of sensorimotor neuropathy (B12 deficiency, Diabetes Mellitus, HIV treated with retroviral medications, thyroid disorders, alcohol abuse, and chronic inflammatory diseases).
10. Co-morbidity anticipated to limit survival to less than 18 months.
11. Patient received an investigational drug/device and/or participated in another clinical investigational study within 60 days before Baseline.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2007-01; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Packman, Study Director — FoldRx Pharmaceuticals, Inc.
Locations (10):
- MGH Neuropathy Laboratory, Boston, Massachusetts, United States
- FLENI-Hepatology and Organ Transplant Dept., Ciudad de Buenos Aires, Buenos Aires, Argentina
- Hospital Universitário Prof. Clementino Fraga Filho-UFRJ, Rio de Janeiro, Southeast, Brazil
- CHU de Bicetre, Le Kremlin-Bicêtre, Île-de-France Region, France
- Universitatsklinikum Munster, Transplant Hepatology, Münster, North Rhine-Westphalia, Germany
- Portugal (2):
  - Serviço de Neurologia-Hospital de Santa Maria, Lisbon, Lisbon District
  - Unidade Clinica de Paramiloidose-Hospital Santo Antonio, Porto, Norte
- Hospital Clinic de Barcelona, Barcelona, Catalonia, Spain
- Umea University Hospital, Umeå, Västerbotten County, Sweden
- Kings College Hospital, London, London, United Kingdom

REFERENCES:
- [Derived] Merlini G, Coelho T, Waddington Cruz M, Li H, Stewart M, Ebede B. Evaluation of Mortality During Long-Term Treatment with Tafamidis for Transthyretin Amyloidosis with Polyneuropathy: Clinical Trial Results up to 8.5 Years. Neurol Ther. 2020 Jun;9(1):105-115. doi: 10.1007/s40120-020-00180-w. Epub 2020 Feb 27. PMID 32107748
- [Derived] Huber P, Flynn A, Sultan MB, Li H, Rill D, Ebede B, Gundapaneni B, Schwartz JH. A comprehensive safety profile of tafamidis in patients with transthyretin amyloid polyneuropathy. Amyloid. 2019 Dec;26(4):203-209. doi: 10.1080/13506129.2019.1643714. Epub 2019 Jul 27. PMID 31353964
- [Derived] Amass L, Li H, Gundapaneni BK, Schwartz JH, Keohane DJ. Influence of baseline neurologic severity on disease progression and the associated disease-modifying effects of tafamidis in patients with transthyretin amyloid polyneuropathy. Orphanet J Rare Dis. 2018 Dec 17;13(1):225. doi: 10.1186/s13023-018-0947-7. PMID 30558645
- [Derived] Gundapaneni BK, Sultan MB, Keohane DJ, Schwartz JH. Tafamidis delays neurological progression comparably across Val30Met and non-Val30Met genotypes in transthyretin familial amyloid polyneuropathy. Eur J Neurol. 2018 Mar;25(3):464-468. doi: 10.1111/ene.13510. Epub 2017 Dec 26. PMID 29115008
- [Derived] Keohane D, Schwartz J, Gundapaneni B, Stewart M, Amass L. Tafamidis delays disease progression in patients with early stage transthyretin familial amyloid polyneuropathy: additional supportive analyses from the pivotal trial. Amyloid. 2017 Mar;24(1):30-36. doi: 10.1080/13506129.2017.1301419. Epub 2017 Apr 10. PMID 28393570
- [Derived] Waddington Cruz M, Amass L, Keohane D, Schwartz J, Li H, Gundapaneni B. Early intervention with tafamidis provides long-term (5.5-year) delay of neurologic progression in transthyretin hereditary amyloid polyneuropathy. Amyloid. 2016 Sep;23(3):178-183. doi: 10.1080/13506129.2016.1207163. Epub 2016 Aug 5. PMID 27494299
- See also: Amyloidosis, Transthyretin-Related — http://www.emedicine.com/med/topic3365.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- Tafamidis: Tafamidis (Fx-1006A) 20 milligram (mg) capsule orally once daily for 18 months.
- Placebo: Placebo, matched to tafamidis (Fx-1006A) 20 mg capsule, orally once daily for 18 months.
Period: Overall Study
Arm/Group | Tafamidis | Placebo
Started | 65 | 63
Completed | 47 | 44
Not Completed | 18 | 19
Not completed — Adverse Event | 4 | 3
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Negative genotype | 0 | 1
Not completed — Liver transplantation | 13 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tafamidis | Placebo | Total
Number analyzed (Participants) | 64 | 61 | 125
Age, Customized [Number; unit: participants] — Out of a total of 128 participants, baseline characteristic (Age) was available for only 125 participants who were included in intent-to-treat (ITT) population.
  participants
    Less than or equal to 65 years | 59 | 58 | 117
    Greater than 65 years | 5 | 3 | 8
Sex: Female, Male [Count of Participants; unit: Participants] — Out of a total of 128 participants, baseline characteristic (Gender) was available for only 125 participants who were included in ITT population.
  Participants
    Female | 32 | 35 | 67
    Male | 32 | 26 | 58

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Response to Treatment as Measured by Neuropathy Impairment Score - Lower Limb (NIS-LL) at Month 18
Description: Response to treatment was indicated by either improvement (decrease from baseline) or stabilization (change from baseline of 0 to less than[<] 2) in NIS-LL score, based on mean of 2 scores in 1 week period. NIS-LL: assessed muscle weakness, reflexes, sensation. Each item scored separately for left, right limbs. Components of muscle weakness scored on 0(normal) to 4(paralysis) scale, higher score=greater weakness. Components of reflexes, sensation scored 0=normal, 1=decreased, or 2=absent. Total NIS-LL score range 0-88, higher score=greater impairment.
Time Frame: Month 18
Population: ITTset:randomized participants received atleast(>=)1 dose of study drug, had >=1 post-baseline efficacy assessment for NIS-LL,Norfolk Quality of Life-Diabetic Neuropathy(QOL-DN) or discontinued study due to death/liver transplant(LT).Last-observation-carried-forward(LOCF) used;participant who discontinued due to death/LT was set non-responder.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tafamidis | Placebo
Number analyzed (Participants) | 64 | 61
percentage of participants | 45.3 [33.1 to 57.5] | 29.5 [18.1 to 41.0]

2. Primary Outcome: Change From Baseline in Norfolk Quality of Life- Diabetic Neuropathy (QOL-DN) Total Quality of Life (TQOL) Score at Month 18
Description: Norfolk QOL-DN: 35-item participant-rated questionnaire used to assess impact of diabetic neuropathy on the quality of life of participants with diabetic neuropathy; Item 1 to 7: related to symptoms and presence of symptom was assessed as 1 and absence was assessed as 0. Item 8-35: related to activities of daily living and scored on a 5-point Likert scale, where 0= no problem and 4= severe problem (except item 32, where -2= much better, 0=about the same, 2=much worse). TQOL= sum of all the items, total possible score range= -2 to 138, where higher score=worse quality of life.
Time Frame: Baseline, Month 18
Population: ITT population included all randomized participants who received at least 1 dose of study medication and had at least 1 post-baseline efficacy assessment for NIS-LL and Norfolk QOL-DN or discontinued study due to death or LT. LOCF method was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tafamidis | Placebo
Number analyzed (Participants) | 64 | 61
units on a scale
  Baseline | 27.3 (24.2) | 30.8 (26.7)
  Change at Month 18 | 2.4 (14.6) | 6.9 (22.9)

3. Secondary Outcome: Change From Baseline in Neuropathy Impairment Score- Lower Limb (NIS-LL) Score at Month 6, 12 and 18
Description: NIS-LL: assessed muscle weakness, reflexes and sensation; scored separately for left and right limbs. Components of muscle weakness (hip and knee flexion, hip and knee extension, ankle dorsiflexors, ankle plantar flexors, toe extensors, toe flexors) are scored on 0(normal) to 4(paralysis) scale, higher score=greater weakness. Components of reflexes (quadriceps femoris, triceps surae) and sensation (touch pressure, pin-prick, vibration, joint position) were scored 0 = normal, 1= decreased, or 2 = absent. Total possible NIS-LL score range 0-88, higher score=greater impairment.
Time Frame: Baseline, Month 6, 12, 18
Population: ITT population included all randomized participants who received at least 1 dose of study medication and had at least 1 post-baseline efficacy assessment for NIS-LL and Norfolk QOL-DN or discontinued study due to death/LT. 'n' = those participants who were evaluable for this measure at given time point for each group respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tafamidis | Placebo
Number analyzed (Participants) | 64 | 61
units on a scale
  Baseline (n=64, 61) | 8.359 (11.399) | 11.445 (13.544)
  Change at Month 6 (n=60, 57) | 1.260 (3.007) | 2.075 (6.407)
  Change at Month 12 (n=49, 50) | 1.005 (3.964) | 4.835 (7.697)
  Change at Month 18 (n=48, 47) | 2.193 (4.372) | 5.402 (8.661)

4. Secondary Outcome: Percentage of Participants With Response to Treatment as Measured by Neuropathy Impairment Score - Lower Limb (NIS-LL) at Month 6 and 12
Description: Response to treatment was indicated by either improvement (decrease from baseline) or stabilization (change from baseline of 0 to <2) in NIS-LL score, based on mean of 2 scores in 1 week period. NIS-LL: assessed muscle weakness, reflexes, sensation. Each item scored separately for left, right limbs. Components of muscle weakness scored on 0 (normal) to 4 (paralysis) scale, higher score=greater weakness. Components of reflexes, sensation scored 0=normal, 1=decreased, or 2=absent. Total NIS-LL score range 0-88, higher score=greater impairment.
Time Frame: Month 6, 12
Population: ITT population included all randomized participants who received at least 1 dose of study medication and had at least 1 post-baseline efficacy assessment for NIS-LL and Norfolk QOL-DN or discontinued study due to death/LT. LOCF method was used; participant who discontinued due to death/LT was set non-responder.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tafamidis | Placebo
Number analyzed (Participants) | 64 | 61
percentage of participants
  Month 6 | 60.9 [49.0 to 72.9] | 54.1 [41.6 to 66.6]
  Month 12 | 54.7 [42.5 to 66.9] | 32.8 [21.0 to 44.6]

5. Secondary Outcome: Change From Baseline in Norfolk Quality of Life - Diabetic Neuropathy (QOL-DN) Total Quality of Life (TQOL) Score at Month 6 and 12
Description: as for outcome 2
Time Frame: Baseline, Month 6, 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tafamidis | Placebo
Number analyzed (Participants) | 64 | 61
units on a scale
  Baseline (n=64, 61) | 27.3 (24.2) | 30.8 (26.7)
  Change at Month 6 (n=60, 57) | 1.2 (15.6) | 0.2 (15.1)
  Change at Month 12 (n=49, 50) | 1.1 (14.7) | 4.6 (19.0)

6. Secondary Outcome: Change From Baseline in Norfolk Quality of Life - Diabetic Neuropathy (QOL-DN) Domain Scores at Month 6, 12 and 18
Description: Norfolk QOL-DN:35-item participant-rated questionnaire to assess impact of DN on QOL; Item 1-7:scored as 1=symptom present, 0=symptom absent. Item 8-35: scored on 5-point Likert scale: 0=no problem, 4=severe problem (except item 32: -2=much better, 0=about same, 2=much worse). Norfolk QOL-DN summarized in 5 domains(score range):physical functioning/large fiber neuropathy(-2 to 58), activities of daily living(ADLs) (0 to 20), symptoms(0 to 32), small fiber neuropathy(0 to 16), autonomic neuropathy(0 to 12); higher score=greater impairment, for each. Total score=-2 to138(higher score=worse QOL).
Time Frame: Baseline, Month 6, 12, 18
Population: ITT population included all randomized participants who received at least 1 dose of study medication and had at least 1 post-baseline efficacy assessment for NIS-LL and Norfolk QOL-DN or discontinued study due to death or LT. 'n' = those participants who were evaluable for this measure at given time points for each group respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tafamidis | Placebo
Number analyzed (Participants) | 64 | 61
units on a scale
  Baseline: physical functioning(n=64,61) | 14.3 (13.8) | 16.6 (14.7)
  Baseline: ADLs(n=64,61) | 1.3 (2.9) | 1.6 (3.8)
  Baseline: symptoms(n=64,61) | 7.2 (5.5) | 7.6 (6.1)
  Baseline: small fiber neuropathy(n=64,61) | 2.7 (3.6) | 3.1 (4.0)
  Baseline: autonomic neuropathy(n=64,61) | 1.9 (2.4) | 2.0 (2.6)
  Change at Month 6: physical functioning(n=60,57) | -0.6 (8.0) | -0.9 (9.8)
  Change at Month 6: ADLs(n=60,57) | 0.4 (1.9) | 0.3 (1.7)
  Change at Month 6: symptoms(n=60,56) | 0.8 (5.5) | 0.2 (4.4)
  Change at Month 6: small fiber neuropathy(n=60,57) | 0.4 (2.2) | 0.5 (2.5)
  Change at Month 6: autonomic neuropathy(n=60,57) | 0.2 (1.8) | 0.0 (1.7)
  Change at Month 12: physical functioning(n=49,50) | -0.9 (7.4) | 0.6 (10.7)
  Change at Month 12: ADLs(n=49,50) | 1.0 (2.4) | 0.7 (3.0)
  Change at Month 12: symptoms(n=49,49) | 0.4 (5.0) | 1.4 (4.5)
  Change at Month 12:small fiber neuropathy(n=49,50) | 0.7 (2.8) | 1.5 (3.1)
  Change at Month 12: autonomic neuropathy(n=49,50) | -0.1 (1.8) | 0.4 (2.8)
  Change at Month 18: physical functioning(n=48,47) | -0.1 (8.5) | 3.0 (14.0)
  Change at Month 18: ADLs(n=48,47) | 1.2 (2.4) | 1.2 (4.2)
  Change at Month 18: symptoms(n=48,47) | -0.1 (4.9) | 1.2 (5.4)
  Change at Month 18:small fiber neuropathy(n=48,47) | 0.8 (2.6) | 1.4 (3.6)
  Change at Month 18: autonomic neuropathy(n=48,47) | 0.2 (1.9) | 0.4 (2.8)

7. Secondary Outcome: Change From Baseline in Summated 7 Score for Large Nerve Fiber Function at Month 6, 12 and 18
Description: Summated 7 score: composite score included five Nerve Conduction Studies (NCS) attributes (peroneal nerve distal motor latency, peroneal nerve compound muscle action potential, peroneal nerve motor conduction velocity, tibial nerve distal motor latency, and sural nerve sensory nerve action potential amplitude) along with Vibration Detection Threshold (VDT) obtained in great toes, and Heart Rate Response to Deep Breathing (HRDB) value. Score was determined through reference to normal values for age, sex and height. Total score range= -26 to 26, where higher score=worse nerve function.
Time Frame: Baseline, Month 6, 12, 18
Population: ITT population included all randomized participants who received at least 1 dose of study medication and had at least 1 post-baseline efficacy assessment for NIS-LL and Norfolk QOL-DN or discontinued study due to death/LT. 'n' = those participants who were evaluable for this measure at given time points for each group respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tafamidis | Placebo
Number analyzed (Participants) | 64 | 61
units on a scale
  Baseline (n=64, 61) | 7.787 (9.063) | 8.718 (8.533)
  Change at Month 6 (n=60, 57) | 0.581 (3.542) | 1.934 (3.846)
  Change at Month 12 (n=48, 50) | 0.833 (3.963) | 2.959 (3.879)
  Change at Month 18 (n=48, 46) | 1.159 (3.853) | 3.333 (4.997)

8. Secondary Outcome: Change From Baseline in Summated 3 Score for Small Nerve Fiber Function at Month 6, 12 and 18
Description: Summated 3 Nerve Tests Small Fiber Normal Deviates Score (NTSFnds) included cooling threshold for the lower limbs, heat pain threshold for the lower limbs and HRDB. Total score range= -11.2 to 11.2, where higher score=worse nerve function.
Time Frame: Baseline, Month 6, 12, 18
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tafamidis | Placebo
Number analyzed (Participants) | 64 | 61
units on a scale
  Baseline (n=64, 61) | 5.514 (4.535) | 5.624 (4.085)
  Change at Month 6 (n=60, 57) | 0.240 (1.679) | 0.716 (2.202)
  Change at Month 12 (n=48, 50) | 0.375 (2.048) | 1.250 (2.010)
  Change at Month 18 (n=48, 46) | 0.290 (2.130) | 1.489 (2.519)

9. Secondary Outcome: Change From Baseline in Modified Body Mass Index (mBMI) at Month 6, 12 and 18
Description: BMI was calculated by weight divided by height squared. mBMI was calculated by multiplying BMI by serum albumin levels to compensate for edema formation associated with malnutrition. A progressive decline in mBMI indicated worsening of disease severity.
Time Frame: Baseline, Month 6, 12, 18
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: (kilogram/square meter)*(gram/liter)
Arm/Group | Tafamidis | Placebo
Number analyzed (Participants) | 64 | 61
(kilogram/square meter)*(gram/liter)
  Baseline (n=64, 61) | 1004.6 (165.2) | 1011.5 (212.9)
  Change at Month 6 (n=60, 56) | 17.1 (68.4) | -29.8 (69.7)
  Change at Month 12 (n=49, 50) | 19.4 (71.8) | -30.8 (74.9)
  Change at Month 18 (n=49, 46) | 37.9 (73.7) | -32.7 (88.6)

10. Secondary Outcome: Percentage of Participants With Stabilized Transthyretin (TTR) Tetramer
Description: TTR tetramer was assessed using a validated immunoturbidimetric assay. The Fraction of Initial (FOI) is the ratio of the measured TTR tetramer concentration after denaturation to the measured TTR tetramer concentration before denaturation. TTR tetramer stabilization is based on the difference between the on-treatment FOI and the baseline FOI expressed as a percentage of the baseline FOI.
Time Frame: Week 8, Month 6, 12, 18
Population: ITT population. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. 'n' = those participants who were evaluable for this measure at given time points for each group respectively.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tafamidis | Placebo
Number analyzed (Participants) | 63 | 60
percentage of participants
  Week 8 (n=63, 60) | 98.4 [95.3 to 100.0] | 6.7 [0.4 to 13.0]
  Month 6 (n= 59, 58) | 100.0 [100.0 to 100.0] | 5.2 [0.0 to 10.9]
  Month 12 (n=48, 50) | 97.9 [93.9 to 100.0] | 2.0 [0.0 to 5.9]
  Month 18 (n=48, 44) | 97.9 [93.9 to 100.0] | 0.0 [0.0 to 0.0]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Tafamidis | Placebo
Serious Adverse Events (participants affected / at risk) | 6/65 | 5/63
Other Adverse Events (participants affected / at risk) | 57/65 | 56/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tafamidis (N=65) | Placebo (N=63)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Conduction disorder (Cardiac disorders) | 1 | 0
Cardiac amyloidosis (Cardiac disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Catheter site phlebitis (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 0
Localised infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Lymphangitis (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1
Burns third degree (Injury, poisoning and procedural complications) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertensive emergency (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tafamidis (N=65) | Placebo (N=63)
Anaemia (Blood and lymphatic system disorders) | 0 | 4
Atrioventricular block first degree (Cardiac disorders) | 2 | 6
Vertigo (Ear and labyrinth disorders) | 3 | 4
Lacrimation decreased (Eye disorders) | 6 | 7
Punctate keratitis (Eye disorders) | 5 | 3
Diarrhoea (Gastrointestinal disorders) | 17 | 11
Nausea (Gastrointestinal disorders) | 8 | 8
Vomiting (Gastrointestinal disorders) | 7 | 7
Constipation (Gastrointestinal disorders) | 4 | 7
Abdominal pain upper (Gastrointestinal disorders) | 8 | 2
Abdominal pain (Gastrointestinal disorders) | 3 | 5
Oedema peripheral (General disorders) | 4 | 8
Fatigue (General disorders) | 0 | 6
Urinary tract infection (Infections and infestations) | 14 | 8
Influenza (Infections and infestations) | 10 | 9
Nasopharyngitis (Infections and infestations) | 9 | 8
Pharyngitis (Infections and infestations) | 4 | 5
Upper respiratory tract infection (Infections and infestations) | 4 | 3
Vaginal infection (Infections and infestations) | 4 | 1
Thermal burn (Injury, poisoning and procedural complications) | 4 | 5
Weight decreased (Investigations) | 3 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 2
Headache (Nervous system disorders) | 10 | 12
Neuralgia (Nervous system disorders) | 2 | 12
Paraesthesia (Nervous system disorders) | 3 | 10
Dizziness (Nervous system disorders) | 2 | 4
Hypoaesthesia (Nervous system disorders) | 1 | 4
Anxiety (Psychiatric disorders) | 4 | 3
Depression (Psychiatric disorders) | 4 | 3
Erectile dysfunction (Reproductive system and breast disorders) | 4 | 4
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 7

LIMITATIONS AND CAVEATS:
Instead of the intended endpoint 'heat pain and cooling threshold', results of 'summated 3 score for small nerve fiber function' were reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.